CLINICAL TRIAL: NCT03624075
Title: Effect of Kinesio Taping on Muscle Force, Pain, Edema, Physical Function and Global Perception of Change of Women With Knee Osteoarthritis: Randomized and Blind Clinical Trial
Brief Title: Effect of Kinesio Taping in Women With Knee Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal do Rio Grande do Norte (Other)
Responsible Party: Principal Investigator, Caio Alano de Almeida Lins, Principal investigator, Universidade Federal do Rio Grande do Norte
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2.577.088
Record Dates: First submitted 2018-06-11; First posted 2018-08-09 (Actual); Last update posted 2020-06-29 (Actual); Status verified 2020-06

CONDITIONS: Kinesio Taping; Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Intervention Model Description: The volunteers will be recruited from the waiting list of the Clinic School of Physiotherapy of the Faculty of Health Sciences of Rio Grande do Norte, as well as the community in general. Initially, a signature will be requested from the TCLE and the next series of personal data. When we are already included, how should participants assess pain, muscular strength, edema and physical function (T0). Then all of them must be allocated to one of the three groups, where due intervention is required for each group. After one session, muscle strength and pain were again assessed (T1) and 72 hours later (T2), all outcomes assessed at time T0 were retested, including the global rating of change.
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- control group (No Intervention): The control group had a protocol of a health education / self-gestation session lasting 60 minutes. This session should include topics such as definition of knee OA, guidance on knee anatomy and physiology, prayer over articulation, rehabilitation and practice of exercises, and as volunteer to receive an educational and self explanatory primer with all the content that is exposed during a lesson .
- Placebo group (Placebo Comparator): The placebo group will simultaneously receive two techniques of applying tensionless KT. The first technique that will be applied is inverted 'Y' on the rectus femoris. In the second technique to be applied, the tape body will be divided lengthwise into four narrow strips. The two pieces intersect the front of the knee. For this application, the volunteer will be positioned in the dorsal position without knee flexion and the tape will be applied by a trained researcher. In the case of bilateral OA, in both techniques of application, the most affected member based on the NPRS score will be the one that will undergo the intervention. All volunteers will remain with the tape for 72 hours.
  Interventions: Other: application of kinesio taping
- intervention group (Experimental): The intervention group will receive the same protocol as the placebo group, differing only in relation to the tension of the bandage. According to Kase et al (2003), the techniques recommend the relief of pain and edema and performance. In the second technique to be applied, the tape body will be divided lengthwise into four narrow strips. The two pieces intersect the front of the knee. For this application, the volunteer will be positioned in the dorsal position without knee flexion and the tape will be applied by a trained researcher. In the case of bilateral OA, in both techniques of application, the most affected member based on the NPRS score will be the one that will undergo the intervention. All volunteers will remain with the tape for 72 hours.
  Interventions: Other: application of kinesio taping

INTERVENTIONS:
Other: application of kinesio taping — application of kinesio taping in the rectus femoris muscle and in the medial and lateral region of the knee
  Arms: Placebo group; intervention group

SUMMARY:
Osteoarthritis (OA) of the knee is a disease characterized mainly by the wear and tear of the articular structures, which affects 6% to 13% of men and 7% to 19% of women, and their prevalence may be increased proportionally with increasing age. Signs and symptoms include pain, joint stiffness and loss of function. In this perspective, kinesio taping (KT) appears as an alternative therapeutic resource for the treatment of this type of patient. However, the current evidence on this technique is limited and conflicting, making its effects on the symptomatology of the disease still uncertain. Thus, the present study will evaluate the effects of KT application on muscle strength, pain, physical function, edema and quality of life of elderly women with knee OA. It will be a randomized, blind clinical trial in which 45 volunteers will be allocated to three groups: G1 (placebo group), G2 (control group) and G3 (intervention group). The G1 will be submitted to the placebo (no tension) application of KT on rectos femoris muscle and knee; the G2 will receive a protocol of a health education activity session lasting 60 minutes and finally the G3 will be submitted to the simultaneous application (with tension) of two KT techniques on rectos femoris muscle and knee. All groups will be evaluated before, immediately after and 72 hours after the application. To measure the variables, the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC), Numerical Pain Rating Scale (NPRS), 6-minute walk test (6MWT), isometric dynamometer, perimetry and global rating of change. Statistical analysis will be done using SPSS® software (Statistical Package Social Science) version 20.0. The Kolmogorov-Smirnov and Levene tests will be applied to evaluate the normality and homogeneity of the data, respectively. Intra and intergroup comparisons will be evaluated using analysis of variance ANOVA of mixed model. In the presence of a significant F, the Benferroni pot-hoc test will be used to identify where the difference occurred. For all statistical analyzes, a significance level of 5% (p <0.05) and 95% confidence interval (95% CI) will be adopted.

ELIGIBILITY:
Inclusion Criteria:

* • Female subjects aged 60 years and over, non-obese (BMI between 18.5 and 24.9 kg / m2), with diagnosis of knee OA according to the criteria of the American College of Rheumatology (Altman et al. , 1986), which are: knee pain most of the day during the last weeks and age greater than 60 years (mandatory criteria), and at least two of the following criteria: stiffness after rest less than 30 minutes, crackle in the affected knee , joint increase of firm consistency, absence of temperature increase and painful hypersensitivity to palpation;

  * Individuals with radiographic signs of degeneration of the knee joint;
  * Individuals with any degree of degeneration according to the Kellgren-Lawrence scale;
  * Individuals with a pain scale above 3 according to NPRS;
  * Stiffness in the knee for at least 6 months prior to screening;
  * Stiffness during the beginning of activities;
  * Intermittent swelling;
  * Never have used KT;
  * Individuals with no history of associated joint disease or systemic rheumatic disease and / or history of surgery in the affected lower limb;
  * Individuals who are not under physiotherapeutic treatment during the intervention;
  * Individuals without neurological, vestibular, visual or auditory deficits that make evaluations impossible.

Exclusion Criteria:

* • Individuals who report pain during the procedure;

  * Individuals who do not complete the treatment time or who do not perform the evaluation procedures correctly, making it impossible to collect any of the data investigated;
  * Individuals with allergy to bandage or cutaneous injury in the region where KT will be applied;
  * Individuals who present hypertensive peak during the evaluations.

Ages: 60 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2018-06-11 (Actual); Primary Completion 2019-03-11 (Actual); Study Completion 2019-06-11 (Actual)

PRIMARY OUTCOMES:
Numerical Pain Rating Scale (NPRS) | Time 0 - baseline
  The primary outcome will pain assessed by the NPRS, whereby participants were asked to choose a number between 0 (no pain) and 10 (worst pain possible). They will instructed to report the level of pain while sitting and rising from a chair.
Numerical Pain Rating Scale (NPRS) | Time 1 - after 10min of the baseline
  The pain of the volunteers will be indirectly measured by the Visual Analogue Scale (VAS), which varies from 0 to 10 (unbearable pain) (SCOTT and HUSKISSON, 1976) . The pain will be measured during the activity of climbing stairs. The patient will be directed to go up and down a staircase with two steps. Initially a volunteer will become familiarized. Volunteers will be guided to perform a normal collective activity (the way they are done in the day). In order to, a voluntary test measure will be used while using an VAS. In VAS, the lower the value, the less the pain sensation realatable by the patient and the higher the value, the greater the pain sensation.
Numerical Pain Rating Scale (NPRS) | Time 2 - after 72 hours of baseline
  The primary outcome will pain assessed by the NPRS, whereby participants were asked to choose a number between 0 (no pain) and 10 (worst pain possible). They will instructed to report the level of pain while sitting and rising from a chair.

SECONDARY OUTCOMES:
Perimetry | Time 0 - baseline
  To perform perimetry, a tape measure will be used to measure the perimeter of the assessed limb. For this, the volunteer will be placed in dorsal decubitus with hip in neutral position, extended knees and relaxed quadriceps. In this position, the evaluator will measure the knee at three specific points: the fold of the popliteal fossa, 5 cm above and 5 cm below. Each level will be evaluated three times and the average of the measurements will be used for analysis.
Perimetry | Time 2 - after 72 hours of baseline
  To perform perimetry, a tape measure will be used to measure the perimeter of the assessed limb. For this, the volunteer will be placed in dorsal decubitus with hip in neutral position, extended knees and relaxed quadriceps. In this position, the evaluator will measure the knee at three specific points: the fold of the popliteal fossa, 5 cm above and 5 cm below. Each level will be evaluated three times and the average of the measurements will be used for analysis.
Quadriceps muscle strength | Time 0 - baseline
  The isometric strength of the femoral quadriceps will evaluated using a hand-held dynamometer (HHD; Nicholas Manual Muscle Tester, Lafayette Instrument Company, Lafayette, Indiana, USA). The participant will placed in the sitting position on a stretcher, with arms crossed over chest. An ankle stabilization belt will placed on the evaluated limb to maintain hip and knee flexion at 90°. The HHD will placed 2 cm proximal to the lateral malleolus midpoint, in the anterior region of the ankle (between the malleoli). Maximum isometric strength will then measured in 5-second knee extensions, with continuous verbal encouragement. Subjects perform one practice trial, rested for 30 s and then carried out the three measured trials, the strongest of which will use for data analysis. The results of all trials [kg] will transformed into Newtons (Strength[N] = strength [kg] x 9.81) and normalized by body mass (Normalized Strength [N/kg] = Strength [N] ÷ Body Mass[kg]).
Quadriceps muscle strength | Time 2 - after 72 hours of baseline
  The isometric strength of the femoral quadriceps will evaluated using a hand-held dynamometer (HHD; Nicholas Manual Muscle Tester, Lafayette Instrument Company, Lafayette, Indiana, USA). The participant will placed in the sitting position on a stretcher, with arms crossed over chest. An ankle stabilization belt will placed on the evaluated limb to maintain hip and knee flexion at 90°. The HHD will placed 2 cm proximal to the lateral malleolus midpoint, in the anterior region of the ankle (between the malleoli). Maximum isometric strength will then measured in 5-second knee extensions, with continuous verbal encouragement. Subjects perform one practice trial, rested for 30 s and then carried out the three measured trials, the strongest of which will use for data analysis. The results of all trials [kg] will transformed into Newtons (Strength[N] = strength [kg] x 9.81) and normalized by body mass (Normalized Strength [N/kg] = Strength [N] ÷ Body Mass[kg]).
Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) | Time 0 - baseline
  Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) is a reliable and validated instrument for the Portuguese language that contains 24 questions divided into three categories: pain (5 questions), rigidity (2 questions) and self-reported physical function (17 questions). The items are evaluated by a Likert scale and each question receives a score ranging from 0 to 96, according to the patient's response. The higher the score obtained, the worse is the severity of the disease (BELLAMY et al., 1988).
Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) | Time 2 - after 72 hours of baseline
  Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) is a reliable and validated instrument for the Portuguese language that contains 24 questions divided into three categories: pain (5 questions), rigidity (2 questions) and self-reported physical function (17 questions). The items are evaluated by a Likert scale and each question receives a score ranging from 0 to 96, according to the patient's response. The higher the score obtained, the worse is the severity of the disease (BELLAMY et al., 1988).
6-minute walk (6MWT) | Time 0 - baseline
  The six-minute walk test (6MWT) will follow the recommendations of the American Thoracic Society (2002). A distance of 30 meters will be demarcated by two cones (one in the initial mark and the other in the final mark). The volunteers will be instructed to walk the greatest number of times the distance marked for six minutes and, at the end of this time, the distance traveled will be measured, in this case, the greater the distance covered, the better the patient's function.
6-minute walk (6MWT) | Time 2 - after 72 hours of baseline
  The six-minute walk test (6MWT) will follow the recommendations of the American Thoracic Society (2002). A distance of 30 meters will be demarcated by two cones (one in the initial mark and the other in the final mark). The volunteers will be instructed to walk the greatest number of times the distance marked for six minutes and, at the end of this time, the distance traveled will be measured, in this case, the greater the distance covered, the better the patient's function.
Global rating of change | Time 2 - after 72 hours of baseline
  This will assessed via the patient global impression of change. The measure is recommended by the Initiative on Methods, Measurement, and Pain Assessment in Clinical Trials group and targets four different domains: pain, function, quality of life, and global condition, measured using a 7-point scale (from 'considerably improved' to 'considerably deteriorated').

CONTACTS AND LOCATIONS:
Locations (1):
- Faculdade de ciências da saúde do trairi - FACISA/UFRN, Santa Cruz, Brazil

REFERENCES:
- [Derived] Pinheiro YT, Barbosa GM, Fialho HRF, Silva CAM, Anunciacao JO, Silva HJA, Souza MC, Lins CAA. Does tension applied in kinesio taping affect pain or function in older women with knee osteoarthritis? A randomised controlled trial. BMJ Open. 2020 Dec 16;10(12):e041121. doi: 10.1136/bmjopen-2020-041121. PMID 33328259